CLINICAL TRIAL: NCT04263259
Title: Efficacy and Mechanisms of Mobile-Delivered Alcohol Attentional Bias Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13419; K01AA023233 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2020-02

CONDITIONS: Alcohol; Harmful Use

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not informed about the nature of the mobile-delivered intervention or their assignment to the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attentional Bias Modification (Experimental): Participants complete attentional bias modification using a dot probe task on a mobile device up to 5 times per day for a 28-day period (80 trials per assessment).
  Interventions: Behavioral: Attentional Bias Modification
- Attentional Bias Control (No Intervention): Participants complete attentional bias assessment-only using a dot probe task on a mobile device up to 5 times per day for a 28-day period (80 trials per assessment).

INTERVENTIONS:
Behavioral: Attentional Bias Modification — Mobile-Delivered Cognitive Retraining Intervention
  Other Names: Cognitive Retraining
  Arms: Attentional Bias Modification

SUMMARY:
This study evaluates the efficacy as well as psychological and neurobiological mechanisms of mobile-delivered alcohol attentional bias modification among heavy drinking adults.

DETAILED DESCRIPTION:
By testing the efficacy and neurobiological mechanisms of behavior change (MOBC) following attentional bias modification among heavy drinking adults, the proposed study has the potential to unify dual process models and neurobiological models of addiction. The cognitive retraining will be delivered via mobile electronic devices to ensure the cost-effectiveness of these procedures, to allow a large amount of retraining to be delivered in an ecologically valid manner, and to facilitate broad dissemination of such procedures if found to be efficacious. Using an intensive longitudinal experimental design, subjects will be randomly assigned into one of 2 groups (attentional bias modification vs. attentional bias control). Ecological momentary assessment (EMA) data will be used to assess changes in cognitive and behavioral measures in situ, and functional magnetic resonance imaging (fMRI) scans before and after cognitive retraining will be used to examine neural changes in specific regions of interest (ROI).

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorders Identification Test greater than or equal to 8
* right-handed

Exclusion Criteria:

* history of treatment for or diagnosis of alcohol use disorder/substance use disorder
* history of brain injury
* for females, currently pregnant
* any MRI safety contraindication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Frequency | 4 weeks
  Number of days of alcohol use during the 4-week ecological momentary assessment period
Alcohol Use Quantity | 4 weeks
  Number of standard drinks per day during the 4-week ecological momentary assessment period
Negative Alcohol-Related Consequences | 4 weeks
  Number negative consequences experienced 4-week ecological momentary assessment period

SECONDARY OUTCOMES:
Attentional Bias to Alcohol | 4 weeks
  Measured with the Alcohol Dot Probe Task
Alcohol Cue-Induced Neural Reward Circuit Activation | 4 weeks
  Regions of interest include ventral tegmental area, dorsal and ventral striatum

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center on Alcoholism, Substance Abuse, & Addictions, Albuquerque, New Mexico
  - Mind Research Network, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers.
Time Frame: Data can be requested from the PI by October 2020
Access Criteria: Data will be shared with qualified scientists who enter a data sharing usage agreement